CLINICAL TRIAL: NCT04095598
Title: Comparative Computed Tomography with Stress Maneuvers for Evaluation of Distal Tibiofibular Syndesmosis Instability in Adults After Acute Ankle Sprain: a Test Accuracy Study
Brief Title: Computed Tomography with Stress Maneuvers for Evaluation of Distal Tibiofibular Syndesmosis Instability (CTMETS)
Acronym: CTMETS
Status: Recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Joao Carlos Rodrigues, Physician, Hospital Israelita Albert Einstein
Other Study IDs: 62100016.5.1001.0071
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Ankle Sprain
Keywords: High ankle sprain; Syndesmotic instability; Computed Tomography; Stress maneuver
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Syndesmotic injured group: The existing index test (ankle CT in neutral position), the new index tests (ankle CT in a stress position with extended-knee; ankle CT in a stress position with flexed-knee), and the reference test (MRI) will be applied. Foot and ankle ability measurement questionnaire (FAAM) will be applied with six months and one year after ankle CT.
  Interventions: Diagnostic Test: Comparative Ankle Tomography with Stress Maneuvers
- Syndesmotic uninjured group: The existing index test (ankle CT in neutral position), the new index tests (ankle CT in a stress position with extended-knee; ankle CT in a stress position with flexed-knee), and the reference test (MRI) will be applied. Foot and ankle ability measurement questionnaire (FAAM) will be applied with six months and one year after ankle CT.
  Interventions: Diagnostic Test: Comparative Ankle Tomography with Stress Maneuvers

INTERVENTIONS:
Diagnostic Test: Comparative Ankle Tomography with Stress Maneuvers — All diagnostic imaging exams and FAAM questionnaire will be applied in a standard way in both groups.

SUMMARY:
The main aim of this study was to investigate which strategy can diagnose more accurately syndesmotic instability among an existing index test (ankle CT in neutral position) and two new add-on index tests (ankle CT in a stress position with extended-knees and ankle CT in a stress position with flexed-knees). This study hypothesized that the two add-on ankle CT with stress maneuvers (CTSM) have a more accurate capability of diagnosing syndesmotic instability than ankle CT in a neutral position (CTNP) alone. The secondary objective is to investigate the participants' disability outcomes by applying the Foot and Ankle Ability Measure questionnaire.

DETAILED DESCRIPTION:
INTRODUCTION:

One specific type of sprain is a high ankle sprain with ligament damage to the distal tibiofibular syndesmosis. A syndesmotic lesion is the leading cause of persistent disability or chronic pain and frequently requires longer recovery times and receives significantly more treatments than low lateral ankle sprains.

The degree of instability in syndesmotic disruption guides the decision to operate or treat conservatively. Clinical examinations, routine radiographs, stress radiographs, computed tomography (CT), and magnetic resonance imaging (MRI) are the available diagnostic tools to decide the correct treatment. Unfortunately, the clinical diagnosis has limited evidence. The best current practice considers that few clinical examination tests have some validity in identifying syndesmotic disruption. The mortise or anteroposterior radiographic view may promptly diagnose frank syndesmotic instability (SI), identifying the widening of the articular space on the injured side relative to the contralateral uninjured side. However, SI may be underdiagnosed when routine radiography shows a healthy articular relationship. Routine radiographs cannot reliably predict syndesmotic injuries. Stress radiographs are inaccurate for evaluating such injuries in a cadaveric model. CTNP is more sensitive than radiography for detecting syndesmotic widening. MRI can be used to visualize and diagnose damaged ligaments with high accuracy.

Notwithstanding, the traditional measurement of the anterior tibiofibular distance (ATFD), obtained by CTNP, has an unsatisfactory area under the receiver operator curve (ROC) performance of 0,58 in diagnosing SI. Despite all these available methods, SI is still challenging to diagnose correctly, and syndesmotic ligament disruption and real SI should be differentiated. CTSM is an alternative approach that could improve the diagnosis of SI. To the investigator's knowledge, the application of CTSM has not been previously described.

METHODS:

This study follows the Standards for Reporting of Diagnostic Accuracy Studies (STARD) guidelines.

Study design:

Diagnostic accuracy-test study.

Study setting:

In partnership with the Department of Orthopedics, the Department of Radiology conducted this study at a tertiary hospital with the approval of the Internal Review Board and the Ethics Committee.

Participant selection and recruitment:

A consecutive sample of individuals with suspected syndesmotic disruption attended at the Foot and Ankle Outpatient Clinic will be referred to the Radiology Department to perform CTNP, CTSM, and MRI. A research assistant (RA) will screen all the participants for eligibility, interview them about their willingness to participate, explain the purposes of the research, and invite those who meet the inclusion criteria to participate. The RA will also describe all study details, answer all questions about objectives, risks, benefits, confidentiality, and read out loud the informed consent form. Individuals who agree to participate will date and sign the informed consent form. The RA will attach a copy of informed consent to the medical record and hand a second copy to the participants. Participants will provide demographic data and complete pre-exams forms before performing image exams. If the participant cannot sign the informed consent form, the RA will provide a verbal explanation of the study. After the verbal consent of the participant, a witness will sign the informed consent form. In addition, RA will record reasons for exclusion or refusal to participate.

CT exam technical parameters:

Aquilion ONE V6 scanner (Toshiba Medical Systems, Tochigi, Japan) with 320 channels will perform all exams using the following technical parameters: a volumetric acquisition, 120 kilovolt, 150 milliampere, 0.5 s rotation time, 0.5 mm slice thickness, 0.25 mm interpolation, 320-detector rows, the field of view (FOV) medium or large, and fine filter for bone. Therefore, the lowest possible irradiation dose will produce images of diagnostic quality. In addition, the feet of the participant will be scanned simultaneously in the same FOV with feet supported on the acrylic board (Medintec, Mogi das Cruzes, Brazil).

MRI exam technical parameters:

A phased array dedicated coil on 1.5-T magnet HDX (GE Healthcare, Milwaukee, USA) will perform all the examinations using the following sequences: sagittal T1-weighted [time repetition (TR)/ echo time (TE), 542/9; number of excitations (NEX), 1; matrix, 320 x 256; thickness, 4 mm; FOV, 10 cm]; sagittal T2-weighted fat-suppressed (3000/39, 2, 384 x 224, 4, 10); axial T2-weighted fat-suppressed (3483/48, 2, 384 x 224, 4, 10); coronal T2-weighted fat-suppressed (3000/39, 2, 384 x 224, 3, 10) and coronal oblique proton density-weighted (2840/35, 2, 384 x 224, 3, 10).

Existing index test (CTNP):

In the neutral phase, the feet will be parallel to each other and perpendicular to the long axis of the legs. The knees will be in an extended position.

New index test (CTSM extended-knees):

In the first stress phase, the feet will be set in external rotation, and voice command will instruct the patient to maintain maximum dorsiflexion to the limit of tolerable pain during image acquisition. The knees will be in an extended position.

New index test (CTSM flexed-knees):

In the second stress phase, the feet will be set in external rotation, and voice command will instruct the patient to maintain maximum dorsiflexion to the limit of tolerable pain during image acquisition. A support pad will keep the knees flexed 30 degrees.

Feasibility assessment:

Investigators will assess feasibility registering all difficulties in performing the maneuvers, including pain exacerbation, motion artifacts, repetition of images, the total duration of the exam, and withdrawal.

CTNP, CTSM extended-knees, and CTSM flexed-knees reading parameters:

Investigators prespecified test positivity cut-off performing measurements of the anterior tibiofibular distance (ATFD) and the posterior tibiofibular distance (PTFD), at 1 cm proximal to the tibial plafond, as described by Elgafy et al. A third measurement will register the smallest distance between the fibula and the tibia, in the plane of the tibiotalar joint, where the CT scan section began to show the whole shape of tibial plafond as described by Ahn et al. All measurements will be obtained in a standardized way in the two ankles of the same individual in the neutral phase and the stress phases. Differences equal to or greater than 1 mm in measures, between the two ankles of the same individual, either in the neutral phase or with stress, will define test positivity cut-off. Although there are no previous studies on stress CT, researchers empirically adopted the 1 mm cut-off point based on a biomechanical study that found considerable changes in the contact area of the tibiotalar joint with lateral talus dislocation of 1 mm or higher.

Reference test (MRI):

The standard protocol will acquire all the ankle MRIs suspected for syndesmotic tear: patients will be scanned with their knees in extension and ankle in a neutral position. Investigators will not scan the unaffected contralateral ankle. The arthroscopic examination is considered the best reference standard for syndesmotic injuries allowing diagnosis and treatment correctly; however, applying this method to the syndesmotic uninjured group would have been difficult to justify ethically. Even a minimally invasive procedure, as the arthroscopic examination, may have complications and is not risk-free. Two studies comparing the accuracy of MRI with arthroscopy concluded that MRI has sensitivity and specificity for evaluating syndesmotic injury close to arthroscopy.

MRI reading parameters:

Investigators prespecified results categories classifying syndesmotic ligaments (anterior inferior tibiofibular, posterior inferior tibiofibular, and interosseous), the lateral collateral ligaments (anterior talofibular, calcaneofibular, and posterior talofibular), and deltoid ligament (superficial and deep layer) as normal, sprain, partial lesion or complete lesion.

Foot and ankle ability measure:

Change in disability will be quantified using the validated version of the Foot and Ankle Ability Measure (FAAM) questionnaire administered at 6 and 12 months after CT. FAAM is a reliable, responsive, and valid tool to evaluate physical activity for various leg, foot, and ankle disorders. A systematic review of the literature identified FAAM as one of the most appropriate patient-assessed tools to quantify functional disabilities in ankle instability.

Blinding and observation bias:

Five groups of individuals will be involved in this study: patients, orthopedics physicians, radiologists physicians, data collectors (research assistants), CTSM and MRI technician performers, and data analysts (statisticians). Blindness will be adopted among them to avoid observation bias. Orthopedists will perform the physical examination blinded to the results of CTSM and MRI. The radiologists will read CTSM blinded to patient identification, physical exam, and laterality of the ankle with the suspected syndesmotic lesion. The radiologists will read MRI blinded to patient identification, physical exam, and CTSM result. The research assistant will collect the questionnaires blinded to the CTSM, MRI, or physical exam results. The technician will perform CTSM blinded to the MRI or physical exam results. Another technician will perform MRI blinded to the CTSM or physical exam results. Researchers will blind the data analysts by labeling the variables with deidentifying terms (such as A and B). Researchers will not communicate participants their group assignments.

Statistical analysis:

Absolute and relative frequencies will describe categorical variables. Median, mean, standard deviation, quartile, minimum and maximum values will describe numerical variables depending on data distribution.

Sensitivity, specificity, AUC, ROC curves, and likelihood ratios (LRs) will be calculated to compare the diagnostic accuracy of the three strategies. The first strategy will test the diagnostic accuracy of the existing index CTNP alone. The second strategy will test the add-on index CTSM extended-knees, and the third will test the add-on index CTSM flexed-knees. "Either positive" rule will be adopted whereby the add-on test is positive if either component test is positive.

Sample size calculation

The most significant sample needed to meet the primary or secondary objective will define the study sample size.

A previous study found the area under de curve (AUC) performance of 0.56 relative to the CT in a neutral position. Assuming as a null hypothesis that the existing CT test has an AUC of 0.56, this study proposes as an alternative hypothesis a new CTSM test with superior accuracy estimated as AUC of 0.80. The full sample size estimated is 39, expecting a 1:2 ratio between groups (13 and 26 cases per group, respectively).

A previous study found that the effect size of the score change paired data in the FAAM sports dimension was 15, the standard deviation of the change in one group was 28, and the other group was 23. Using a two-sample paired t-test to compare the changes in FAAM score, the full sample size estimation is 111, expecting a 1:2 ratio between groups (37 and 74 cases per group, respectively). Accounting for a possible loss of 20% during follow-up, investigators intend to include 133 participants in the study. The same methodology applied for the activity of daily life (ADL) domain in the FAAM score found a full sample size of 60 participants.

The sample size of 133 for the sports domain contemplates the ADL domain and the AUC sample calculation of 60 and 39, respectively.

ELIGIBILITY:
Inclusion criteria:

* Adults older than 18 years;
* One episode of an ankle sprain;
* Sprain episode occurred up to 3 weeks prior;
* Positive orthopedic evaluation for suspected syndesmotic injury.

Exclusion criteria

* Bilateral ankle sprain;
* Previous ankle surgery;
* Ankle fractures and dislocations (except avulsion fractures in ligamentous insertions or fracture of the posterior malleolus related to syndesmotic injury);
* Congenital or acquired ankle deformities;
* Infection, inflammatory, or neuropathic ankle arthropathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients seen at the foot and ankle outpatient clinic of a tertiary hospital with an orthopedic clinical diagnosis of syndesmotic lesion will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Tibiofibular distance | Through the study completion, a average of three years
  Measurements of the tibiofibular distance

SECONDARY OUTCOMES:
Foot and Ankle Ability Measurement | Change from 6 months to 12 months
  Functional scale with two subscales (daily life activity and sport) reported separately. The scale range for each subscale varies from the lowest score value (zero) to the highest value (100) in percentage. Higher scores represent a better outcome for both subscales.
Interobserver CT agreement reliability | Through the study completion, a average of three years
  Intraclass correlation coefficient for CT continuous data
Interobserver MRI agreement reliability | Through the study completion, a average of three years
  Kappa coefficient for MRI categorical data

CONTACTS AND LOCATIONS:
Overall Officials: João Carlos Rodrigues, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelista Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerber JP, Williams GN, Scoville CR, Arciero RA, Taylor DC. Persistent disability associated with ankle sprains: a prospective examination of an athletic population. Foot Ankle Int. 1998 Oct;19(10):653-60. doi: 10.1177/107110079801901002. PMID 9801078
- [Background] Boytim MJ, Fischer DA, Neumann L. Syndesmotic ankle sprains. Am J Sports Med. 1991 May-Jun;19(3):294-8. doi: 10.1177/036354659101900315. PMID 1907807
- [Background] van Dijk CN, Longo UG, Loppini M, Florio P, Maltese L, Ciuffreda M, Denaro V. Conservative and surgical management of acute isolated syndesmotic injuries: ESSKA-AFAS consensus and guidelines. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1217-27. doi: 10.1007/s00167-016-4017-1. Epub 2016 Feb 4. PMID 26846658
- [Background] van Dijk CN, Longo UG, Loppini M, Florio P, Maltese L, Ciuffreda M, Denaro V. Classification and diagnosis of acute isolated syndesmotic injuries: ESSKA-AFAS consensus and guidelines. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1200-16. doi: 10.1007/s00167-015-3942-8. Epub 2015 Dec 24. PMID 26704800
- [Background] Krahenbuhl N, Weinberg MW, Davidson NP, Mills MK, Hintermann B, Saltzman CL, Barg A. Imaging in syndesmotic injury: a systematic literature review. Skeletal Radiol. 2018 May;47(5):631-648. doi: 10.1007/s00256-017-2823-2. Epub 2017 Nov 30. PMID 29188345
- [Background] Beumer A, Valstar ER, Garling EH, van Leeuwen WJ, Sikma W, Niesing R, Ranstam J, Swierstra BA. External rotation stress imaging in syndesmotic injuries of the ankle: comparison of lateral radiography and radiostereometry in a cadaveric model. Acta Orthop Scand. 2003 Apr;74(2):201-5. doi: 10.1080/00016470310013969. PMID 12807330
- [Background] Oae K, Takao M, Naito K, Uchio Y, Kono T, Ishida J, Ochi M. Injury of the tibiofibular syndesmosis: value of MR imaging for diagnosis. Radiology. 2003 Apr;227(1):155-61. doi: 10.1148/radiol.2271011865. Epub 2003 Feb 28. PMID 12616009
- [Background] Ebraheim NA, Lu J, Yang H, Mekhail AO, Yeasting RA. Radiographic and CT evaluation of tibiofibular syndesmotic diastasis: a cadaver study. Foot Ankle Int. 1997 Nov;18(11):693-8. doi: 10.1177/107110079701801103. PMID 9391813
- [Background] Ahn TK, Choi SM, Kim JY, Lee WC. Isolated Syndesmosis Diastasis: Computed Tomography Scan Assessment With Arthroscopic Correlation. Arthroscopy. 2017 Apr;33(4):828-834. doi: 10.1016/j.arthro.2017.01.009. Epub 2017 Feb 23. PMID 28237080
- [Background] Cohen JF, Korevaar DA, Altman DG, Bruns DE, Gatsonis CA, Hooft L, Irwig L, Levine D, Reitsma JB, de Vet HC, Bossuyt PM. STARD 2015 guidelines for reporting diagnostic accuracy studies: explanation and elaboration. BMJ Open. 2016 Nov 14;6(11):e012799. doi: 10.1136/bmjopen-2016-012799. PMID 28137831
- [Background] Elgafy H, Semaan HB, Blessinger B, Wassef A, Ebraheim NA. Computed tomography of normal distal tibiofibular syndesmosis. Skeletal Radiol. 2010 Jun;39(6):559-64. doi: 10.1007/s00256-009-0809-4. Epub 2009 Oct 15. PMID 19830423
- [Background] Ramsey PL, Hamilton W. Changes in tibiotalar area of contact caused by lateral talar shift. J Bone Joint Surg Am. 1976 Apr;58(3):356-7. PMID 1262367
- [Background] Teramoto A, Kura H, Uchiyama E, Suzuki D, Yamashita T. Three-dimensional analysis of ankle instability after tibiofibular syndesmosis injuries: a biomechanical experimental study. Am J Sports Med. 2008 Feb;36(2):348-52. doi: 10.1177/0363546507308235. Epub 2007 Oct 16. PMID 17940143
- [Background] Eechaute C, Vaes P, Van Aerschot L, Asman S, Duquet W. The clinimetric qualities of patient-assessed instruments for measuring chronic ankle instability: a systematic review. BMC Musculoskelet Disord. 2007 Jan 18;8:6. doi: 10.1186/1471-2474-8-6. PMID 17233912
- [Background] Moreira TS, Magalhaes Lde C, Silva RD, Martin RL, Resende MA. Translation, cross-cultural adaptation and validity of the Brazilian version of the Foot and Ankle Ability Measure questionnaire. Disabil Rehabil. 2016 Dec;38(25):2479-90. doi: 10.3109/09638288.2015.1137979. Epub 2016 Feb 15. PMID 26878102
- [Background] Vogl TJ, Hochmuth K, Diebold T, Lubrich J, Hofmann R, Stockle U, Sollner O, Bisson S, Sudkamp N, Maeurer J, Haas N, Felix R. Magnetic resonance imaging in the diagnosis of acute injured distal tibiofibular syndesmosis. Invest Radiol. 1997 Jul;32(7):401-9. doi: 10.1097/00004424-199707000-00006. PMID 9228606
- [Derived] Rodrigues JC, Santos ALG, Prado MP, Alloza JFM, Masagao RA, Rosemberg LA, Barros DDCS, Castro ADAE, Demange MK, Lenza M, Ferretti M. Comparative CT with stress manoeuvres for diagnosing distal isolated tibiofibular syndesmotic injury in acute ankle sprain: a protocol for an accuracy- test prospective study. BMJ Open. 2020 Sep 3;10(9):e037239. doi: 10.1136/bmjopen-2020-037239. PMID 32883728